CLINICAL TRIAL: NCT05443282
Title: Serum Prolidase Activity in Primary Ovarian Insufficiency
Brief Title: Ovarian Reserve and Matrix Metalloproteinases
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Esin Merve Erol Koç, Medical Doctor, Ankara City Hospital Bilkent
Other Study IDs: E1-20-1189
Record Dates: First submitted 2022-06-24; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Oxidative Stress; Ovarian Insufficiency, Primary; Ovarian Failure, Premature
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the serum samples of peripheral venous blood obtained from antecubital vein were used to analyze prolidase, proline and hydroxyproline levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POI group (Study group): * The study group included 68 women with POI.
  * The POI cases had been diagnosed as idiopathic POI.
  * The POI diagnosis was based on the presence of amenorrhea before the age of 40, increased serum FSH level higher than 40 mIU/ml, and decreased estradiol levels lesser than 50 pg/mL.
  Interventions: Diagnostic Test: Prolidase Level; Diagnostic Test: Follicle Stimulating Hormone Level; Diagnostic Test: Estradiol Level; Diagnostic Test: Proline Level; Diagnostic Test: Hydroxyproline Level; Diagnostic Test: Anti-mullerian Hormone Level; Diagnostic Test: Antral Follicle Count; Diagnostic Test: Prolactine Level; Diagnostic Test: Thyroid Stimulating Hormone Level
- Normally menstruating women (Control group): * Control group consisted of 65 healthy, regularly menstruating women.
  * The women were at the age of lesser than 40 years old.
  * The women were recruited consecutively from those that applied to outpatient clinics to get counselling for family planning.
  Interventions: Diagnostic Test: Prolidase Level; Diagnostic Test: Follicle Stimulating Hormone Level; Diagnostic Test: Estradiol Level; Diagnostic Test: Proline Level; Diagnostic Test: Hydroxyproline Level; Diagnostic Test: Anti-mullerian Hormone Level; Diagnostic Test: Antral Follicle Count; Diagnostic Test: Prolactine Level; Diagnostic Test: Thyroid Stimulating Hormone Level

INTERVENTIONS:
Diagnostic Test: Prolidase Level — Measurement of venous blood serum level of prolidase enzyme level by ELISA method.
Diagnostic Test: Follicle Stimulating Hormone Level — Measurement of venous blood serum level of follicle stimulating hormone level.
Diagnostic Test: Estradiol Level — Measurement of venous blood serum level of estradiol hormone level.
Diagnostic Test: Proline Level — Measurement of venous blood serum level of proline level.
Diagnostic Test: Hydroxyproline Level — Measurement of venous blood serum level of hydroxyproline level.
Diagnostic Test: Anti-mullerian Hormone Level — Measurement of venous blood serum level of anti-mullerian hormone level.
Diagnostic Test: Antral Follicle Count — Ultrasonographic evaluation of antral follicle count to determine ovarian reserve.
Diagnostic Test: Prolactine Level — Measurement of venous blood serum prolactine hormone level.
Diagnostic Test: Thyroid Stimulating Hormone Level — Measurement of venous blood serum thyroid stimulating hormone level.

SUMMARY:
Primary Ovarian Insufficiency (POI) is dysfunction of ovaries before 40 years of age. It has been reported that genetic factors, endocrine disorders, previous pelvic surgeries, chemotherapy and radiotherapy, and autoimmune mechanisms play a role in 10%, however the etiology has not been clarified in 90% of the cases. Oxidative stress and autoimmunity has been shown to be responsible in the etiopathogenesis of POI. Prolidase is an imidodipeptidase. Prolidase was shown to be related with oxidative stress and autoimmune diseases in previous studies. In addition, it is thought that the level of prolidase plays a role both in the etiopathogenesis and progression of diseases. This study aims to investigate the level of prolidase enzyme in women with POI.

DETAILED DESCRIPTION:
Primary Ovarian Insufficiency (POI) is dysfunction of ovaries before 40 years of age. It has been reported that genetic factors, endocrine disorders, previous pelvic surgeries, chemotherapy and radiotherapy, and autoimmune mechanisms play a role in 10%, however the etiology has not been clarified in 90% of the cases that are diagnosed as idiopathic POI. Recent studies concentrated on the role of immune mechanisms in idiopathic POI. Prolidase is a matrix metalloproteinase that plays a role in various metabolic processes and is responsible for the destruction of dipeptides containing proline and hydroxyproline. The prolidase has been shown to be related with oxidative stress and autoimmune diseases in previous studies. Prolidase was shown to be a diagnostic and prognostic value in a number of diseases. Proline and hydroxyproline are metabolites produced through the prolidase activity. Proline itself is also considered as a kind of metabolic stress indicator. On the other hand, free proline in the medium is known to inhibit the prolidase enzyme activity. Therefore, simultaneous measurement of proline and hydroxyproline levels in the medium enables to more accurately calculate the prolidase activity. This study aim to analyze the prolidase level in POI patients compared to healthy menstruating women. Besides the prolidase activity, we also aim to measure proline and hydroxyproline levels in order to provide the calibration for accurate results in terms of prolidase activity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of POI for study group
* Regularly menstruating women for control group
* Normally developed secondary sexual characteristics

Exclusion Criteria:

* Cardiovascular diseases including hypertension
* Type 1 or type 2 diabetes mellitus
* Morbid obesity
* Primary adrenal insufficiency
* Uterine fibroids
* Thyroid dysfunctions including Hashimoto thyroiditis and Grave's disease
* Hepatic dysfunctions
* Renal insufficiency
* Genetic disorders in chromosome constitution or karyotype analysis including monosomy X, trisomy X and gene mutations as BMP15, FMR I, POFIB, and GDF9
* Neurologic diseases
* Psychiatric disorders
* Autoimmune diseases or syndromes including Addison's disease, autoimmune syndromes, scleroderma, Sjogren's syndrome, myasthenia gravis, inflammatory bowel diseases, multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus and familial Mediterranean fever
* History of any malignancy
* History of exposure to chemotherapeutic agents or radiotherapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POI means early cessation of menses, thus it is a disease diagnosed in only females.
Study Population: Study population includes a total of 133 participants. The study group consists of 68 women with the diagnosis of idiopathic POI, and the control group consists of 65 normally menstruating women.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Serum prolidase level | 10 minutes
  Units per liter

SECONDARY OUTCOMES:
Serum proline level | 10 minutes
  Micromole per liter
Serum hydroxyproline level | 10 minutes
  Micromole per liter

CONTACTS AND LOCATIONS:
Overall Officials: Esin Merve Erol Koç, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD are available which may be shared in necessary conditions.

REFERENCES:
- [Result] Committee opinion no. 605: primary ovarian insufficiency in adolescents and young women. Obstet Gynecol. 2014 Jul;124(1):193-197. doi: 10.1097/01.AOG.0000451757.51964.98. PMID 24945456
- [Result] Szeliga A, Calik-Ksepka A, Maciejewska-Jeske M, Grymowicz M, Smolarczyk K, Kostrzak A, Smolarczyk R, Rudnicka E, Meczekalski B. Autoimmune Diseases in Patients with Premature Ovarian Insufficiency-Our Current State of Knowledge. Int J Mol Sci. 2021 Mar 5;22(5):2594. doi: 10.3390/ijms22052594. PMID 33807517
- [Result] Rafique S, Sterling EW, Nelson LM. A new approach to primary ovarian insufficiency. Obstet Gynecol Clin North Am. 2012 Dec;39(4):567-86. doi: 10.1016/j.ogc.2012.09.007. PMID 23182561
- [Result] Namiduru ES. Prolidase. Bratisl Lek Listy. 2016;117(8):480-5. doi: 10.4149/bll_2016_093. PMID 27546702
- [Result] Zhou F, Shi LB, Zhang SY. Ovarian Fibrosis: A Phenomenon of Concern. Chin Med J (Engl). 2017 Feb 5;130(3):365-371. doi: 10.4103/0366-6999.198931. PMID 28139522
- [Result] Hart RJ. Physiological Aspects of Female Fertility: Role of the Environment, Modern Lifestyle, and Genetics. Physiol Rev. 2016 Jul;96(3):873-909. doi: 10.1152/physrev.00023.2015. PMID 27252278
- [Result] Kitchener RL, Grunden AM. Prolidase function in proline metabolism and its medical and biotechnological applications. J Appl Microbiol. 2012 Aug;113(2):233-47. doi: 10.1111/j.1365-2672.2012.05310.x. Epub 2012 May 10. PMID 22512465
- [Result] Practice Committee of the American Society for Reproductive Medicine. Testing and interpreting measures of ovarian reserve: a committee opinion. Fertil Steril. 2015 Mar;103(3):e9-e17. doi: 10.1016/j.fertnstert.2014.12.093. Epub 2015 Jan 10. PMID 25585505
- [Result] Myara I, Charpentier C, Lemonnier A. Optimal conditions for prolidase assay by proline colorimetric determination: application to iminodipeptiduria. Clin Chim Acta. 1982 Oct 27;125(2):193-205. doi: 10.1016/0009-8981(82)90196-6. PMID 7139961
- [Result] Huang Y, Hu C, Ye H, Luo R, Fu X, Li X, Huang J, Chen W, Zheng Y. Inflamm-Aging: A New Mechanism Affecting Premature Ovarian Insufficiency. J Immunol Res. 2019 Jan 2;2019:8069898. doi: 10.1155/2019/8069898. eCollection 2019. PMID 30719458
- [Result] Bakalov VK, Anasti JN, Calis KA, Vanderhoof VH, Premkumar A, Chen S, Furmaniak J, Smith BR, Merino MJ, Nelson LM. Autoimmune oophoritis as a mechanism of follicular dysfunction in women with 46,XX spontaneous premature ovarian failure. Fertil Steril. 2005 Oct;84(4):958-65. doi: 10.1016/j.fertnstert.2005.04.060. PMID 16213850
- [Result] Luborsky J. Ovarian autoimmune disease and ovarian autoantibodies. J Womens Health Gend Based Med. 2002 Sep;11(7):585-99. doi: 10.1089/152460902760360540. PMID 12396892
- [Result] Goswami D, Conway GS. Premature ovarian failure. Hum Reprod Update. 2005 Jul-Aug;11(4):391-410. doi: 10.1093/humupd/dmi012. Epub 2005 May 26. PMID 15919682
- [Result] Carp HJ, Selmi C, Shoenfeld Y. The autoimmune bases of infertility and pregnancy loss. J Autoimmun. 2012 May;38(2-3):J266-74. doi: 10.1016/j.jaut.2011.11.016. Epub 2012 Jan 27. PMID 22284905
- [Result] La Marca A, Broekmans FJ, Volpe A, Fauser BC, Macklon NS; ESHRE Special Interest Group for Reproductive Endocrinology--AMH Round Table. Anti-Mullerian hormone (AMH): what do we still need to know? Hum Reprod. 2009 Sep;24(9):2264-75. doi: 10.1093/humrep/dep210. Epub 2009 Jun 11. PMID 19520713